CLINICAL TRIAL: NCT06729827
Title: Non-invasive PREDIctive Hemodynamic Continuous moniToring vs Standard Intermittent Blood Pressure and Post-spinal hypotensION During Elective Cesarean Section: a Randomized Clinical Trial
Brief Title: Predictive Hemodynamic Monitoring During Elective Cesarean Section
Acronym: PREDICTION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FRASSANITO LUCIANO, Dr, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5508
Record Dates: First submitted 2024-12-07; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related; Cesarean Section Complications; Hypotension on Induction; Anesthesia Complication
Keywords: Spinal induced hypotension; cesarean section; hypotension nprediction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Predictive monitoring - HPI (Experimental): In the HPI-group the patients will be treated with a bolus of norepinephrine 5 mcg each time that HPI is 85 or higher.
  Interventions: Device: Hypotension prediction Index - HPI
- Control group (No Intervention): In the control group a rescue bolus of norepinephrine 5 mcg will be administered by the anesthesia care provider whenever MAP decreases below 65 mmHg.

INTERVENTIONS:
Device: Hypotension prediction Index - HPI — Patients in the HPI group, in addition to standard monitoring, will have hemodynamic monitoring using HemoSphere (Edwards Lifesciences, Irvine, CA) with ClearSight non-invasive hemodynamic monitoring and with the HPI software enabled.
  The patients will be treated with a bolus of norepinephrine 5 mcg each time that HPI is 85 or higher.
  Arms: Predictive monitoring - HPI

SUMMARY:
Single shot spinal anesthesia (SA) is the most commonly used technique for Caesarean section (CS) .

SA is associated with maternal hypotension (Post Spinal Hypotension - PSH) often accompanied by nausea, vomiting, bradycardia and fetal acidosis.

Preventive administration of vasopressors is widely used to counterbalance hypotension.

Routine prophylactic infusion of phenilephrine and norepinephrine raises concerns for unnecessary treatment, reactive hypertension, baroreceptor-mediated bradycardia, and effects on fetal acidosis.

Non-invasive continuous measurement of arterial pressure using a finger cuff is well established. Hypotension Prediction Index - HPI is an algorithm that could predict the onset of hypotension in working on invasive and non-invasive arterial waveform signal.

The aim of this prospective randomized study is to compare the amount of PSH during elective caesarean section among two groups of patients receiving standard intermittent hemodynamic monitoring versus continuous ClearSight-HPI monitoring. The primary hypothesis is that hemodynamic management HPI-guided reduces the incidence, entity and duration of post-spinal hypotension, defined as mean arterial pressure (MAP) lower than 65 mmHg lasting more than one minute.

Our secondary aim was to study the impact of maternal PSH during CS on foetal outcome evaluated by comparing neonatal Apgar scores at 1 and 5 minutes after birth, and umbilical cord arterial and venous pH in the two groups.

DETAILED DESCRIPTION:
Caesarean section (CS) is one of the most commonly performed operations worldwide, with 1 in 5 women (21.1%) currently giving birth through this route.

The introduction of neuraxial techniques determined an improved safety, better postoperative analgesia, reduction in hemorrhage, higher Apgar scores in the neonate and a more participative birth experience.

Single shot spinal anesthesia (SA) is the most commonly used technique because it provides rapid onset, effective and reliable anesthesia.

SA induces a sympathetic block that almost inevitably produces maternal hypotension (Post Spinal Hypotension - PSH) often accompanied by nausea, vomiting and bradycardia. Sustained PSH may lead to decreased utero-placental blood flow and fetal acidosis. For this reason, the optimal management of hypotension in this setting has become one of the most active areas of research in obstetric anesthesia. In particular, preventive administration of vasopressors directly counter arteriolar vasodilation and decreased systemic vascular resistance and, by maintaining vascular tone in venous and splanchnic vessels, increases venous return and cardiac filling.

Although proactive vasopressor administration is now considered the strategy of choice for PSH, the ideal drug, dose, and mode of delivery have been debated. Studies comparing prophylactic phenylephrine infusions and rescue boluse doses have shown conflicting results. Routine prophylactic vasopressor infusion raises concerns for unnecessary or even inappropriate treatment, particularly when hypotension is unlikely to develop (50%). In other words, half of the patients, those not experiencing spinal-induced hypotension, may be exposed to unnecessary vasopressor infusion potentially developing adverse effects such as hypertension, tachycardia, Takotsubo cardiomyopathy, ventricular arrhythmias. Prophylactic phenylephrine infusions have gained favor, as recommended by the latest published international consensus statement. On the other hand, continuous vasopressors infusions may be detrimental to hemodynamic homeostasis, potentially resulting in reactive hypertension or precipitating a baroreceptor-mediated bradycardia, which in turn may result in reduced maternal CO: indeed, cardiac output decreases significantly with increasing phenylephrine rate. Norepinephrine prophylaxis is gaining popularity in clinical practice because of less bradycardia and higher maternal CO compared with phenylephrine prophylaxis. Nevertheless, concerns about an effect of norepinephrine on fetal acidosis were raised by several authors: lower umbilical pH using continuous infusion of vasopressors probably result from placental transfer and stimulation of foetal metabolism.

Several authors suggest individual patient characteristics, for example body mass index (BMI) and pre-operative anxiety, as predictors of hypotension, with mixed results. Cardiovascular variables have been studied as early indicators of maternal hypotension including baseline heart rate (HR), changes in HR variability after the SA, cerebral near infrared spectroscopy and cardiac ultrasound parameters. International guidelines suggest that there is an increased risk of maternal hypotension if the baseline HR is high or increased after the spinal local anesthetic injection.

Non-invasive measurement of the arterial pressure using a finger cuff (ClearSight, Edwards Lifesciences, Irvine, USA) is well established.

The Hypotension Prediction Index - HPI (Edwards Lifesciences, Irvine, USA) is an algorithm based on the complex analysis of features in high fidelity arterial pressure waveform recordings developed to observe subtle signs that could predict the onset of hypotension in surgical and intensive care unit patients. HPI is a unitless number that ranges from 1 to 100, and as the number increases, the likelihood of a hypotensive event (defined as a mean arterial pressure [MAP] of <65 mmHg for more than 1 minute) occurring in the near future increases. In a validation study on HPI conducted in non-obstetric patients under general anesthesia, the algorithm, at its optimal value, predicted hypotension with both sensitivity and specificity of 86% (95% CI, 86% to 86%) 5 minutes before the event. The performance of HPI in awake pregnant patients has been studied: it provides an accurate real time and continuous prediction of impending intraoperative hypotension before its occurrence with an acceptable agreement between MAP measured by ClearSight and conventional NIBP monitoring.

Patients in the control group will undergo standard monitoring (Life Scope TR, Nihon Kohden Co, Tokyo, Japan) included a 5-lead electrocardiogram, pulse oximetry and NIBP with an upper arm cuff.

Patients in the HPI group, in addition to standard monitoring, will have hemodynamic monitoring using HemoSphere (Edwards Lifesciences, Irvine, CA) with ClearSight non-invasive hemodynamic monitoring and with the HPI software enabled. The clocks of the HemoSphere and Life Scope TR will be synchronized (degree of precision: +/- 1 second).

After arriving at the operating theatre, each patient will be laid on the operating table with a comfortable medical pad and an obstetric wedge will be placed under the right buttock.

The ClearSight system will be applied to the left hand of the patient and continuous hemodynamic monitoring will start. Each patient will have a resting base-line measurement for 5 min, and the average arterial pressure value will be recorded as the baseline value.

All data from the HemoSphere monitor (Edwards Lifesciences, Irvine, CA) will be downloaded as follows: HPI, cardiac output, cardiac index, MAP, systolic arterial pressure, diastolic arterial pressure, HR, stroke volume, stroke volume variation, pulse pressure variation, contractility and dynamic arterial elastance. All downloaded data consist in 20-second interval averaged data points.

Anesthetic management A large bore i.v. catheter will be inserted in a forearm vein, and Cefazolin 2 g, Metoclopramide 10 mg and Omeprazole 40 mg will be administered. SA will be performed in sitting position after local infiltration with 2% Lidocaine, using a 25-G Whitacre spinal needle, preferentially at the L3-4 vertebral interspace, with hyperbaric 0.5% bupivacaine plus sufentanil 5 mcg and morphine 100 mcg. The bupivacaine dose will be adjusted for height: 8 mg for patients < 160 cm tall, 9 mg for patients between 160 and 170 cm, and 10 mg for those >170 cm. The patients will be then positioned supine with the wedge under the right buttock. Rapid fluid administration with Ringer Lactate solution (to administer 7 mL/kg as co-load) will be started until delivery. After delivery, fluid management will be left to discretion of the attending anesthesiologist. The level of sensory block will be assessed using a sterile 27-G Whitacre needle, aiming for a level of anesthesia at T4. After delivery, Oxytocin will be administered to facilitate uterine contraction.

Hypotension treatment In the control group a rescue bolus of norepinephrine 5 mcg will be administered by the anesthesia care provider whenever MAP decreases below 65 mmHg.

In the HPI-group the patients will be treated with a bolus of norepinephrine 5 mcg each time that HPI is 85 or higher.

Bradycardia (defined as a HR <45 bpm or HR<60 bpm plus hypotension) will be treated by atropine 0.5 mg or ephedrine 5 mg.

Hypertensive episodes (MAP > 110 mmHg) will be registered.

Fetal wellbeing Samples of umbilical arterial (UA) and umbilical venous (UV) blood will be collected from a double-clamped segment of umbilical cord. We will collect Apgar scores at 1 and 5min after delivery.

Statistic plan The data will be described in their demographic and clinical characteristics through the application of descriptive statistics. The qualitative variables will be described using tables of absolute frequencies and percentages; the continuous quantitative variables will be presented as a median and interquartile range or as a mean and standard deviation when normally distributed; while the non-normal variables will be presented as minimum, maximum and median values.

In the two groups of patients, the hypotensive events, defined as a MAP lower than 65mmHg for > 1 minute (and the severe hypotensive events as having a MAP lower than 60 and 55 mmHg), will be analyzed in terms of frequency and absolute duration and, to estimate their severity, as the ratio between the area under the 65 mmHg threshold and the total length, expressed in minutes, of intraoperative monitoring using the TWA-MAP method.

The Chi-squared test will be used to compare the two incidences. The t-student test for independent samples will be used to evaluate statistically significant differences among the patients' demographic and anthropometric characteristics. The Shapiro-Wilk test will be used to assess the normality of data distribution, while the sd test will be used to verify the equality of the variance. The Mann-Whitney test will be used for independent samples to compare the data that are not normally distributed.

Regarding the assessment of the secondary outcomes, the investigators will report the relative risks with 95% confidence intervals and p-values based on either the chi square or Fisher's exact test, as more appropriate according to the frequencies expected and detected.

A p-value <0.05 will be considered statistically significant. All of the analysis will be performed through the STATA IC 15.1 (Stata Corp) for Windows, Microsoft Excel, Matlab (The MathWorks Inc., Natick, MA, USA) and the Acumen Analytics software (Edwards Lifesciences, Irvine, CA).

ELIGIBILITY:
Inclusion Criteria:

* Full term pregnancy
* Elective cesarean section under spinal anesthesia
* Age > 18 years

Exclusion Criteria:

* refusal to participate to the study
* preeclampsia
* cardiovascular diseases
* neuromuscular disease;
* emergent or urgent cesarean delivery;
* coagulopathies;
* contraindications to spinal anesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 102 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
AUC-MAP<65 mmHg 20 min | In the first 20 min after Spinal Anesthesia
  Area under the curve (AUC) for Mean Arterial Pressure < 65 mmHg.

SECONDARY OUTCOMES:
Fetal wellbeing - 1 | At the birth of the fetus
  Umbelical cord arterial pH, venous pH and base excess,
Fetal wellbeing - 2 | After 5 min from the birth of the fetus
  APGAR score performed by neonatologist
TWA-MAP < 65 mmHg | At the end of the surgery.
  time weighted average (TWA) MAP < 65 mmHg in the total length, expressed in minutes, of intraoperative monitoring.

OTHER OUTCOMES:
Total fluids and vasopressor use | At the end of the surgery.
  Total amount of fluids and vasopressors used during the surgery.
Maternal side effects | At 2 hours after surgery.
  Incidence of maternal side effects

REFERENCES:
- [Background] Knutzen L, Svirko E, Impey L. The significance of base deficit in acidemic term neonates. Am J Obstet Gynecol. 2015 Sep;213(3):373.e1-7. doi: 10.1016/j.ajog.2015.03.051. Epub 2015 Mar 28. PMID 25827502
- [Result] Betran AP, Ye J, Moller AB, Souza JP, Zhang J. Trends and projections of caesarean section rates: global and regional estimates. BMJ Glob Health. 2021 Jun;6(6):e005671. doi: 10.1136/bmjgh-2021-005671. PMID 34130991
- [Result] Bamber JH, Lucas DN, Plaat F, Russell R. Obstetric anaesthetic practice in the UK: a descriptive analysis of the National Obstetric Anaesthetic Database 2009-14. Br J Anaesth. 2020 Oct;125(4):580-587. doi: 10.1016/j.bja.2020.06.053. Epub 2020 Jul 28. PMID 32736825
- [Result] Mercier FJ, Auge M, Hoffmann C, Fischer C, Le Gouez A. Maternal hypotension during spinal anesthesia for caesarean delivery. Minerva Anestesiol. 2013 Jan;79(1):62-73. Epub 2012 Nov 18. PMID 23135692
- [Result] Fratelli N, Prefumo F, Andrico S, Lorandi A, Recupero D, Tomasoni G, Frusca T. Effects of epidural analgesia on uterine artery Doppler in labour. Br J Anaesth. 2011 Feb;106(2):221-4. doi: 10.1093/bja/aeq317. Epub 2010 Nov 24. PMID 21106576
- [Result] Valentin M, Ducarme G, Ceccaldi PF, Bougeois B, Luton D. Uterine artery, umbilical, and fetal cerebral Doppler velocities after epidural analgesia during labor. Int J Gynaecol Obstet. 2012 Aug;118(2):145-8. doi: 10.1016/j.ijgo.2012.03.034. Epub 2012 May 19. PMID 22613492
- [Result] Antoine C, Young BK. Fetal lactic acidosis with epidural anesthesia. Am J Obstet Gynecol. 1982 Jan 1;142(1):55-9. doi: 10.1016/s0002-9378(16)32284-0. PMID 7055172
- [Result] Dyer RA, Biccard BM. Ephedrine for spinal hypotension during elective caesarean section: the final nail in the coffin? Acta Anaesthesiol Scand. 2012 Aug;56(7):807-9. doi: 10.1111/j.1399-6576.2012.02719.x. No abstract available. PMID 22780437
- [Result] Doherty A, Ohashi Y, Downey K, Carvalho JC. Phenylephrine infusion versus bolus regimens during cesarean delivery under spinal anesthesia: a double-blind randomized clinical trial to assess hemodynamic changes. Anesth Analg. 2012 Dec;115(6):1343-50. doi: 10.1213/ANE.0b013e31826ac3db. Epub 2012 Sep 25. PMID 23011562
- [Result] Siddik-Sayyid SM, Taha SK, Kanazi GE, Aouad MT. A randomized controlled trial of variable rate phenylephrine infusion with rescue phenylephrine boluses versus rescue boluses alone on physician interventions during spinal anesthesia for elective cesarean delivery. Anesth Analg. 2014 Mar;118(3):611-8. doi: 10.1213/01.ane.0000437731.60260.ce. PMID 24299932
- [Result] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Result] Stewart A, Fernando R, McDonald S, Hignett R, Jones T, Columb M. The dose-dependent effects of phenylephrine for elective cesarean delivery under spinal anesthesia. Anesth Analg. 2010 Nov;111(5):1230-7. doi: 10.1213/ANE.0b013e3181f2eae1. Epub 2010 Sep 14. PMID 20841418
- [Result] Ngan Kee WD, Lee SW, Ng FF, Tan PE, Khaw KS. Randomized double-blinded comparison of norepinephrine and phenylephrine for maintenance of blood pressure during spinal anesthesia for cesarean delivery. Anesthesiology. 2015 Apr;122(4):736-45. doi: 10.1097/ALN.0000000000000601. PMID 25635593
- [Result] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Result] Davies SJ, Vistisen ST, Jian Z, Hatib F, Scheeren TWL. Ability of an Arterial Waveform Analysis-Derived Hypotension Prediction Index to Predict Future Hypotensive Events in Surgical Patients. Anesth Analg. 2020 Feb;130(2):352-359. doi: 10.1213/ANE.0000000000004121. PMID 30896602
- [Result] Akkermans J, Diepeveen M, Ganzevoort W, van Montfrans GA, Westerhof BE, Wolf H. Continuous non-invasive blood pressure monitoring, a validation study of Nexfin in a pregnant population. Hypertens Pregnancy. 2009 May;28(2):230-42. doi: 10.1080/10641950802601260. PMID 19437233
- [Result] Maheshwari K, Buddi S, Jian Z, Settels J, Shimada T, Cohen B, Sessler DI, Hatib F. Performance of the Hypotension Prediction Index with non-invasive arterial pressure waveforms in non-cardiac surgical patients. J Clin Monit Comput. 2021 Feb;35(1):71-78. doi: 10.1007/s10877-020-00463-5. Epub 2020 Jan 27. PMID 31989416
- [Result] Juri T, Suehiro K, Kimura A, Mukai A, Tanaka K, Yamada T, Mori T, Nishikawa K. Impact of non-invasive continuous blood pressure monitoring on maternal hypotension during cesarean delivery: a randomized-controlled study. J Anesth. 2018 Dec;32(6):822-830. doi: 10.1007/s00540-018-2560-2. Epub 2018 Sep 28. PMID 30267340
- [Result] Frassanito L, Sonnino C, Piersanti A, Zanfini BA, Catarci S, Giuri PP, Scorzoni M, Gonnella GL, Antonelli M, Draisci G. Performance of the Hypotension Prediction Index With Noninvasive Arterial Pressure Waveforms in Awake Cesarean Delivery Patients Under Spinal Anesthesia. Anesth Analg. 2022 Mar 1;134(3):633-643. doi: 10.1213/ANE.0000000000005754. PMID 34591796
- [Result] Noto A, Sanfilippo F, De Salvo G, Crimi C, Benedetto F, Watson X, Cecconi M, David A. Noninvasive continuous arterial pressure monitoring with Clearsight during awake carotid endarterectomy: A prospective observational study. Eur J Anaesthesiol. 2019 Feb;36(2):144-152. doi: 10.1097/EJA.0000000000000938. PMID 30562226
- [Result] Kouz K, Weidemann F, Naebian A, Lohr A, Bergholz A, Thomsen KK, Krause L, Petzoldt M, Moll-Khosrawi P, Sessler DI, Flick M, Saugel B. Continuous Finger-cuff versus Intermittent Oscillometric Arterial Pressure Monitoring and Hypotension during Induction of Anesthesia and Noncardiac Surgery: The DETECT Randomized Trial. Anesthesiology. 2023 Sep 1;139(3):298-308. doi: 10.1097/ALN.0000000000004629. PMID 37265355
- [Result] Caesarean birth. London: National Institute for Health and Care Excellence (NICE); 2021 Mar 31. Available from http://www.ncbi.nlm.nih.gov/books/NBK569570/ PMID 33877751